CLINICAL TRIAL: NCT00436631
Title: Internet Administration of the Modified Atkins Diet for Adults With Intractable Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Eric Kossoff, Professor, Neurology, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00008471
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Epilepsy
Keywords: epilepsy; seizures; intractable; ketosis; ketogenic; diet
MeSH Terms: conditions — Epilepsy; Seizures; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diet (Experimental)
  Interventions: Behavioral: Dietary management of seizures

INTERVENTIONS:
Behavioral: Dietary management of seizures — Using the high-fat, low carbohydrate modified Atkins diet - 15 grams per day initially. This is a 3-month study of this diet.

SUMMARY:
This is a prospective, open-label (no control or blind) study to continue to determine whether the modified Atkins diet reduces seizures, creates ketosis, and is well tolerated in adults (not children) with epilepsy. This study will enroll and manage patients via email, phone, and fax and without dietitian involvement (primary difference from previous studies). It is a 3 month study.

DETAILED DESCRIPTION:
Patients will have contacted either Dr. Kossoff or Dr. Cervenka either via referral or self-referral.

Inclusion: over 18 years of age, at least weekly seizures (or 4 per month), tried at least 2 medications for your seizures, have email and fax access, are not very underweight or have high cholesterol, have not had status epilepticus (seizure lasting over 30 minutes) in the past 6 months, and have not tried the Atkins diet before or the ketogenic diet within the past year. All patients will need to have a local primary care doctor or neurologist willing to be available in case of emergencies. You and your local physician both need to speak and write in English and patients MUST be in the United States to participate. The patient (NOT a caregiver) must be the person to email the investigators - a family member cannot be the contact person.

If the patient agrees, we will send and they will fax back within 2 weeks:

1. Signed consent
2. Signed note from their neurologist/primary care provider (attached)
3. 6 months of medical records to confirm their qualification
4. 3-day food record (can be emailed by the patient)
5. Labs (CBC, CMP, fasting lipid profile, urine calcium, urine creatinine, urine hcG (if female) (form attached)

After that, we will send information on how to do the diet via email, they will maintain monthly calendars, and after 3 months we will decide if the diet is helpful. After that time point, they can continue it on their own with periodic followup with either us or their local neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients must consent for themselves (NOT a family member doing this).
* Patients need to be willing to perform the induction phase of the diet.
* Patients must have access to an email account and fax machine.
* Persisting, countable seizures (> 1 per week or 4 times per month) despite previous treatment with two or more antiepileptic drugs.
* Patients with coronary heart disease, cerebrovascular disease, peripheral vascular disease, atherosclerosis, prior myocardial infarctions, or renal dysfunction will be excluded.

Exclusion Criteria:

* Patients previously exposed to the Atkins diet (for more than one week) will be excluded.
* Patients who had tried the ketogenic diet within the past year will be excluded.
* Patients with non-epileptic seizures (pseudoseizures) will be excluded.
* Patients that are pregnant or become pregnant during the study will be excluded.
* Patients must have a local English-speaking neurologist or primary care provider willing to sign a form stating they are available for any emergencies, considering some patients may be a far distance away.
* Patients must live in the United States.
* Patients must not have a history of status epilepticus within the past 6 months.
* Patients with a BMI that is below 18.5 will be excluded.
* Patients must speak and write in English.
* Patients must be from the United States.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | 3 months

SECONDARY OUTCOMES:
Tolerability (ability to create and maintain ketosis), cholesterol, weight | 3 months
Ability to follow instructions via email (and maintain ketosis and seizure control when achieved). | 3 months
Ketosis (measured by urine) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kossoff EH, McGrogan JR, Bluml RM, Pillas DJ, Rubenstein JE, Vining EP. A modified Atkins diet is effective for the treatment of intractable pediatric epilepsy. Epilepsia. 2006 Feb;47(2):421-4. doi: 10.1111/j.1528-1167.2006.00438.x. PMID 16499770
- [Background] Kossoff EH, Rowley H, Sinha SR, Vining EP. A prospective study of the modified Atkins diet for intractable epilepsy in adults. Epilepsia. 2008 Feb;49(2):316-9. doi: 10.1111/j.1528-1167.2007.01256.x. Epub 2007 Oct 5. PMID 17919301
- See also: Information about this approach from a parent — http://www.atkinsforseizures.com